CLINICAL TRIAL: NCT05961319
Title: Smart Home Technologies for Assessing and Monitoring Frailty in Older Adults
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: Alberta Health services (Other); Glenrose Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00131722
Record Dates: First submitted 2023-06-26; First posted 2023-07-27 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Frailty; Frailty Syndrome; Frail Elderly Syndrome; Pre-Frailty; Healthy; Healthy Aging; Aging Problems; Aging Disorder
Keywords: Frail; Frailty; Pre-Frail; Assessment; Monitoring; Home; House; Smart; Technology; Technological; Sensors; Tracking
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Utilizing Smart Home Monitoring System in a Simulated Home Environment (in Hospital): The project involves recruiting participants who will reside in a simulated condo environment within the Glenrose Rehabilitation Hospital. These participants will be remotely monitored using various sensors, including ones that track their interactions with appliances and furniture, smart biomechanics devices that assess their physical balance and strength, and a positioning system. By collecting and analyzing data from these sensors, the project aims to gain insights into the participants' daily activities, functional abilities, physical condition, and spatial behaviour.
  Interventions: Device: Smart-Home Monitoring

INTERVENTIONS:
Device: Smart-Home Monitoring — During the study, various sensors will be employed to capture participant interactions with appliances and furniture. These sensors may include:
  Interaction Sensors: These sensors are designed to recognize users' interactions with appliances and furniture within the smart environment.
  Smart Biomechanics Devices: Devices such as a Fitbit device an internet of Things grip Dynamometer will be utilized to assess physical balance and strength.
  Positioning System using Ultra-Wide Band (UWB) Technology: This positioning system leverages UWB technology, enabling furniture-level accuracies in interpreting self-care activities.
  As participants engage with different elements of the smart environment, these sensors will collect data. Additionally, participants will be recorded via video to further enhance the observational data captured during the study.

SUMMARY:
This project aims to address the impact of frailty on older adults, particularly its connection to cognitive impairments such as dementia. By identifying frailty in its early stages, interventions can be designed to slow down the progression of cognitive decline. To achieve this, the project plans to develop a reliable at-home monitoring system that can accurately track frailty in older adults with mild cognitive impairment or dementia. By utilizing cutting-edge technologies such as high-precision indoor positioning and home-installed sensors, referred to as zero-effort technologies (ZETs), the system will collect continuous sensor data, which will be analyzed to identify indicators of frailty.

DETAILED DESCRIPTION:
This project is centred around addressing the impact of frailty on older adults and its correlation with cognitive impairments, particularly dementia. The aim is to develop an effective and non-intrusive at-home monitoring system that can accurately track frailty in older adults with mild cognitive impairment or dementia. By identifying frailty in its early stages, interventions can be designed to slow down the progression of cognitive decline and improve the overall well-being of older adults.

To achieve this, the project plans to leverage cutting-edge technologies such as high-precision indoor positioning and home-installed sensors, collectively referred to as zero-effort technologies (ZETs). These technologies require minimal user effort and will provide a continuous stream of sensor data. The collected data will be systematically analyzed to identify indicators of frailty, allowing for early detection and intervention. Importantly, the project recognizes the significance of engaging older adults, caregivers, and healthcare professionals throughout the development process. Their attitudes, beliefs, and perceptions will be taken into consideration to ensure that the monitoring system is meaningful, beneficial, and respects user privacy.

By involving older adults and caregivers in the early stages, the project aims to create a monitoring system that can be seamlessly integrated into the lives of older adults dealing with frailty and cognitive impairments. The goal is to provide an affordable and efficient solution that can be implemented within the comfort and familiarity of their own homes. The continuous tracking of frailty data will enable healthcare professionals and caregivers to deliver timely interventions and support, thereby potentially slowing down the cognitive decline experienced by older adults.

Through the combination of advanced technologies and a user-centred approach, the project intends to bridge the gap between frailty and cognitive impairments in older adults. By identifying frailty at an early stage and tailoring interventions accordingly, personalized and targeted support can be provided to improve the quality of life for older adults with mild cognitive impairment or dementia. Ultimately, the project aims to contribute to the development of effective strategies for managing frailty and cognitive decline, benefiting both older adults and their caregivers, as well as clinicians.

ELIGIBILITY:
Inclusion Criteria:

* In-patients at the Glenrose Rehabilitation Hospital (GRH) and GRH' visitors or staff (e.g. patients' caregivers, relatives, friends of older adults in-patient or staff at the GRH who are interested in participating) who are 65 years old or older
* For in-patients who are pre-frail or frail according to the scale used at the GRH (can be equivalent to Fried's scale pre-frail/frail (score = 1 - 4). For GRH's visitors or staff, are robust according to Fried's Frail Scale (score=0) as per the definition in (Fried, 2001)
* With or without some level of cognitive impairment (Standardized mini-mental state examination (MMSE) of 21 to 30 ("mild" (24-21) to "could be normal" (25-30)) or the equivalent in the screening tool.
* Have a cognitive ability to interact with the frailty sensors (i.e. scale, dynamometer, smart speaker).
* Have a functional vision and hearing with or without aides (glasses/hearing aids) to be able to interact with furniture and sensors at the ILS and to fill out questionnaires.
* Have functional upper extremity function to be able to interact with furniture and sensors at the ILS.
* Be able to walk independently 15 meters with or without a walking aid.
* If taking antidepressants or narcotics, participants have no changes in the medication for at least 3 months

Exclusion Criteria:

* Those with a history of Parkinson's disease or other movement disorders or stroke.

Justification: Movement disorders causing tremors will affect data collection by the sensors

* Those who were taking Sinemet or Aricept
* Older adults who have Influenza, long Covid-19 or another virus that affect their performance
* Unable to count, speak (name objects and say numbers) or comprehend simple instructions in English
* Have severe cardiac or respiratory diseases that prevent them to perform vigorous activities
* Using supplemental oxygen (i.e., must be able to breathe with room air)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Older aged adults (60+ years old), with or without frailty, and with or without mild cognitive impairment (MCI).
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Slowness (Mobility) | through study completion, within a total average of 2 hours
  15 Foot Walk / 5 Metres, Timed. The sensors and the camera will record the participants' data during this time.
Weight (lbs, Kgs) | through study completion, within a total average of 2 hours
  Weight taken using an internet of things scale
Exhaustion | through study completion, within a total average of 2 hours
  Smart speaker delivered two questions from the Center for Epidemiological Studies-Depression (CES-D) scale (7. I felt that everything I did was an Effort, 20. I could not get "going."). The sensors and the camera will record the participants' data during this time.
Strength - Handgrip | through study completion, within a total average of 2 hours
  Using a internet of things dynanometer, force will be assessed (3 times each hand - 30 seconds of rest between measurements) and to release it. The sensors and the camera will record the participants' data during this time.
Activity | through study completion, within a total average of 2 hours
  The participant is asked to complete two tasks from the Performance Assessment of Self-Care Skills (PASS - Clinic) Version 4.1. This will involve a simulated version of carrying garbage, and sweeping the floors. The sensors and the camera will record the participants' data during this time.
Meal Preparation | through study completion, within a total average of 2 hours
  Participants will be asked to prepare a simple sandwich using the kitchen elements.The sensors and the camera will record the participants' data during this time.
Observe Free Activity | through study completion, within a total average of 2 hours
  During the data collection, participants will be given 5 minutes to do whatever activity they want. The sensors and the camera will record the participants' data during this time.
Qualitative Interviews Regarding Technology | Through study completion, within a total average of 2 hours
  Qualitative Interview (Based on the Unified Theory of Acceptance and Use of Technology (UTAUT) constructs)

CONTACTS AND LOCATIONS:
Overall Officials: Jim Raso, MASc, Study Chair — Alberta Health services
Locations (2):
- Canada (2):
  - Glenrose Rehabilitation Hospital, Edmonton, Alberta
  - Corbett Hall, University of Alberta, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lewinsohn PM, Seeley JR, Roberts RE, Allen NB. Center for Epidemiologic Studies Depression Scale (CES-D) as a screening instrument for depression among community-residing older adults. Psychol Aging. 1997 Jun;12(2):277-87. doi: 10.1037//0882-7974.12.2.277. PMID 9189988
- [Background] Chisholm D, Toto P, Raina K, Holm M, Rogers J. Evaluating capacity to live independently and safely in the community: Performance Assessment of Self-care Skills. Br J Occup Ther. 2014 Feb;77(2):59-63. doi: 10.4276/030802214X13916969447038. PMID 25298616
- [Background] Venkatesh, V., Morris, M. G., Davis, G. B., & Davis, F. D. (2003). User Acceptance of Information Technology: Toward a Unified View. MIS Quarterly, 27(3), 425-478. https://doi.org/10.2307/30036540
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204